CLINICAL TRIAL: NCT07190963
Title: Detection of Concussion and Recovery Study
Brief Title: MindRhythm Detection of Concussion and Recovery Study
Acronym: DISCOVERY
Status: Recruiting | Type: Observational
Sponsor: MindRhythm, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mTBI-002MR
Record Dates: First submitted 2025-07-07; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: mTBI - Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Concussed: An individual who is diagnosed or suspected of having a mTBI or concussion
- Normal: An individual who has not been diagnosed or suspected of having a mTBI or concussion within one preceding year

SUMMARY:
This study is designed to observe HeadPulse data in concussed subjects that may have experienced a concussion via an injury down to the age of 4. Sports teams are the focus of this study because therein lies inherent potential risk for concussion. This observational study will further confirm the data previously collected in professional athletes to further validate that the HeadPulse can be used as a digital biometric to objectively indicate when a concussed brain remains concussed despite a subject feeling no symptoms has extreme value. This study is intended to support the development of a device to objectively determine when it is safe to return to play or normal activity based on the output of the digital biometric.

ELIGIBILITY:
Inclusion Criteria: An individual who has been diagnosed with or suspected to have a concussion or mTBI.

-

Exclusion Criteria: open wounds on the head. Pregnant women due to unexpected risks. Subjects under the age of 4.

-

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have experienced a mTBI/concussion compared to a cohort of cohort of neurologically normal individuals who have not experienced diagnosed or undiagnosed concussion or head trauma within the last 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2027-01-28 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is measurement and aggregate evaluation of the time course of HeadPulse abnormalities and the proportion of subjects who later worsen following clearance to return to activities. | Subject data will be acquired for approximately 30 days from subject enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- MindRhythm Incorporated, Cupertino, California, United States